CLINICAL TRIAL: NCT06513689
Title: Pleural Fluid Proteomics From Patients With Pleural Infection Shows Signatures of Diverse Neutrophilic Responses: The Oxford Pleural Infection Endotyping Study (TORPIDS 2)
Brief Title: The Oxford Pleural Infection Endotyping Study
Acronym: TORPIDS-2
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: R74885/RE001
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-06

CONDITIONS: Pleural Infection; Pleural Diseases; Pleural Effusion; Pleural Empyema; Pleural Infection Bacterial; Pleural Infections and Inflammations
Keywords: pleural; pleural infection; respiratory; neutrophils
MeSH Terms: conditions — Pleural Diseases; Pleural Effusion; Empyema, Pleural; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Acellular pleural fluid specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolment: All samples were collect at patient enrolment for the PILOT study (PMID: 32675200, ISRCTN 50236700)

SUMMARY:
Pleural infection is a severe disease with increasing incidence worldwide. The subphenotypes of pleural infection remain unknown.We designed a study to endotype the disease and assess the association between patient phenotype, microbiology and clinical outcome.

We subjected 80 pleural fluid samples to unlabelled mass spectrometry.

Pathway analysis of the differentially expressed proteins identified the neutrophil degranulation, glycolysis, pentose phosphate pathway, and the liver and retinoid X receptors (LXR-RXR) activation. Higher neutrophil degranulation was associated with increased glycolysis and pentose phosphate activation.

Pleural infection patients exhibit proteomic signatures indicating diverse responses of neutrophil mediated immunity, glycolysis, and pentose phosphate activation.

DETAILED DESCRIPTION:
Pleural infection is a common and severe disease with increasing incidence worldwide. The endotypes of pleural infection remain unknown. A better understanding of patient variation in underlying biological response to infection may lead to improved treatments and clinical outcomes. We designed a study with the aim to endotype the disease and assess the association between patient phenotype, microbiology and clinical outcome.

We subjected 80 pleural fluid samples from the PILOT study, a prospective study on pleural infection, to unlabelled mass spectrometry. Proteins were retained if they were detected in at least 50% of the samples resulting in a total of 449 proteins. Unsupervised hierarchical clustering and UMAP analyses were used to cluster samples, Spearman and exact Fischer's methods were used for correlation assessment and protein expression was correlated with clinical outcomes.

UMAP plotting separated the samples in to two different and distinct cohorts. Pathway analysis of the differentially expressed proteins identified neutrophil degranulation, glycolysis, the pentose phosphate pathway, and the liver and retinoid X receptors (LXR-RXR) activation. Higher neutrophil degranulation was associated with increased glycolysis and pentose phosphate activation. Specimens dominated by Streptococcus Pneumoniae exhibited high neutrophil degranulation. Increased activity of the LXR-RXR pathway was associated with better survival.

Pleural infection patients exhibit proteomic signatures indicating diverse responses of neutrophil mediated immunity, glycolysis, and pentose phosphate activation which were associated with microbiology. Therapeutic targeting the LXR-XRX pathway with agonists may improve survival.

ELIGIBILITY:
Samples collected for the PILOT clinical trial (DOI: 10.1183/13993003.00130-2020) used for the TORPIDS-2 study.

Patients were included if they had a clinical presentation consistent with pleural infection and any of the following criteria: 1. pleural fluid that was macroscopically purulent; or 2. pleural fluid that was positive on culture for bacterial infection; or 3. pleural fluid that demonstrated bacteria on Gram staining; or 4. pleural fluid with a pH ≤7.2 (measured by blood gas analyser) or low glucose level (≤3 mmol·L-1 or ≤55 mg·dL-1) in a patient with clinical evidence of infection; or 5. contrast-enhanced computed tomography (CT) evidence of pleural infection (consolidation of underlying lung with enhancing pleural collection) in a patient with clinical evidence of infection, alongside exclusion of other sources of infection. Evidence of infection was assessed by the recruiting physician on the basis of fever, an elevated peripheral blood white-cell count, or elevated serum inflammatory markers such as C-reactive protein (CRP). Study exclusion criteria were as follows: 1. age <18 years; 2. no pleural fluid available for analysis; 3. previous pneumonectomy on the side of pleural infection; and 4. expected survival of <3 months due to co-morbid disease, as judged by the recruiting physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with evidence of pleural infection
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Pleural infection endotypes | 12 months
  Discovery of pleural infection biological endotypes
Association between endotypes and microbiology | 12 months
  Investigate the association between pleural infection endotypes and microbiology
Association between endotypes and one-year survival | 12 months
  Investigate the association between pleural infection endotypes and one-year survival

SECONDARY OUTCOMES:
Association between endotypes and need for surgical treatment | 12 months
  Investigate the association between pleural infection endotypes and need for surgical treatment
Association between levels of pleural fluid plasminogen and neutrophil elastase | 12 months
  Investigate the association between pleural fluid plasminogen and neutrophil elastase protein levels

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Pleural Translational Research, Nuffield Department of Medicine, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised and non-identifiable data could be shared with other researchers. The mass spectrometry data are deposited in PRIDE to share with other researchers.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] "Prospective validation of the RAPID clinical risk prediction score in adult patients with pleural infection: the PILOT study." John P. Corcoran, Ioannis Psallidas, Stephen Gerry, Francesco Piccolo, Coenraad F. Koegelenberg, Tarek Saba, Cyrus Daneshvar, Ian Fairbairn, Richard Heinink, Alex West, Andrew E. Stanton, Jayne Holme, Jack A. Kastelik, Henry Steer, Nicola J. Downer, Mohammed Haris, Emma H. Baker, Caroline F. Everett, Justin Pepperell, Thomas Bewick, Lonny Yarmus, Fabien Maldonado, Burhan Khan, Alan Hart-Thomas, Georgina Hands, Geoffrey Warwick, Duneesha De Fonseka, Maged Hassan, Mohammed Munavvar, Anur Guhan, Mitra Shahidi, Zara Pogson, Lee Dowson, Natalia D. Popowicz, Judith Saba, Neil R. Ward, Rob J. Hallifax, Melissa Dobson, Rachel Shaw, Emma L. Hedley, Assunta Sabia, Barbara Robinson, Gary S. Collins, Helen E. Davies, Ly-Mee Yu, Robert F. Miller, Nick A. Maskell and Najib M. Rahman. Eur Respir J 2020; 56: 2000130. Eur Respir J. 2020 Dec 17;56(6):2050130. doi: 10.1183/13993003.50130-2020. Print 2020 Dec. No abstract available. PMID 33334780